CLINICAL TRIAL: NCT06510621
Title: The Preliminary Application of Socket-shield Technique in Orthodontic Extraction and Fixed Orthodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Yuhang Zhang, Director, Department of Stomatology, Principal Investigator, Clinical Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 201827
Record Dates: First submitted 2024-07-08; First posted 2024-07-19 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Immediate Dental Implant Loading
Keywords: Socket-Shield Technique; Bone preservation; First premolar extraction; Orthodontics
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Socket-Shield Technique (Experimental): Cut the tooth crown; divided along the long axis; trim the socket shield. Finally, the socket-shield was removed by minimally invasive forceps when the adjacent tooth moved proximate to the shield during the process of closing orthodontic gap.
  Interventions: Procedure: Socket-Shield Technique
- non-Socket-Shield Technique (No Intervention): A high-speed turbine was used to cut the tooth crown 1.5-2 mm from the buccal gingival margin. The tooth was then divided along the long axis, approximately 2 mm from the buccal side. The palatal roots were removed using minimally invasive elevation and extraction forceps. Next, the buccal socket-shield was trimmed to approximately 4-6 mm in height (1 mm from the buccal gingival margin), 3-4 mm in width, and 1-1.5 mm in thickness. The trimming process required with clear visualization of the shield and calibration by periodontal probe. Finally, the socket-shield was removed immediately

INTERVENTIONS:
Procedure: Socket-Shield Technique — A high-speed turbine was used to cut the tooth crown 1.5-2 mm from the buccal gingival margin. The tooth was then divided along the long axis, approximately 2 mm from the buccal side(Figure 1c, 1d). The palatal roots were removed using minimally invasive elevation and extraction forceps. Next, the buccal socket-shield was trimmed to approximately 4-6 mm in height (1 mm from the buccal gingival margin)[18], 3-4 mm in width, and 1-1.5 mm in thickness[19,20]. The trimming process required with clear visualization of the shield and calibration by periodontal probe. Finally, the socket-shield was removed by minimally invasive forceps when the adjacent tooth moved proximate to the shield during the process of closing orthodontic gap.
  Arms: Socket-Shield Technique

SUMMARY:
Background This study was conducted to investigate the clinical efficacy of Socket-Shield Technique on the first premolar bone preservation in Orthodontic Extraction Treatment.

Methods patients were underwent Orthodontic Extraction Treatment in the First Affiliated Hospital of Guangzhou Medical University were enrolled. Extracted teeth were paired and randomly allocated into two groups: test group (Socket-Shield Technique) and control group. Cone beam computerized tomography were utilized to access the horizontal resorption and vertical resorption at 1mm, 3mm and 5mm from a reference plane of alveolar crest, as well as tooth movement rate at four time-points: before tooth extraction (T0), three months after tooth extraction (T1), the juncture socket-shield was removed (T2) and three months after socket-shield removal (T3).

DETAILED DESCRIPTION:
2.1 Participants This study was conducted following the Declaration of Helsinki, the Consolidates Standards of Reporting Trials (CONSORT), and the Good Clinical Practice (GCP) guideline. The protocol was reviewed and approved by the Ethics Committee of the First Affiliated Hospital of Guangzhou Medical University (Approval No. 2018-27). All patients were informed and agreed to provide informed consent and their data for further analysis and publication. Additionally, for minors participating in the study, informed consent was obtained from a parent or legal guardian.

Patients were included in the study if they reached all of the following criteria: (1) had an orthodontic treatment plan involving the extraction of symmetrical left and right first premolars; (2) had maxillary protrusion or bimaxillary protrusion with crowding within 4mm; (3) had permanent dentition; (4) had good oral hygiene and had no periodontitis; and (5) agreed to the orthodontic extraction treatment plan and signed the treatment informed consent form and the experimental informed consent form.

The study exclusion criteria were as follows: (1) underlying diseases such as hypertension, heart disease, diabetes, osteoporosis, or hyperthyroidism; (2) infection in the extraction area; (3) dental root caries in the extraction area; (4) gingival recession on the buccal aspect of the extraction area; (5) refused to undergo SST treatments; and (6) pregnancy or lactation.

2.2 Surgical procedure Test Group (SST): A high-speed turbine was used to cut the tooth crown 1.5-2 mm from the buccal gingival margin (Figure 1a, 1b). The tooth was then divided along the long axis, approximately 2 mm from the buccal side(Figure 1c, 1d). The palatal roots were removed using minimally invasive elevation and extraction forceps. Next, the buccal socket-shield was trimmed to approximately 4-6 mm in height (1 mm from the buccal gingival margin)[18], 3-4 mm in width, and 1-1.5 mm in thickness. The trimming process required with clear visualization of the shield and calibration by periodontal probe. Finally, the socket-shield was removed by minimally invasive forceps when the adjacent tooth moved proximate to the shield during the process of closing orthodontic gap.

Control Group (non-SST): The same technique was used to cut the crown, divide the root, remove the palatal root, trim the socket-shield, and extract the shield immediately .

After the tooth extraction, patients were prescribed clindamycin and ibuprofen sustained-release capsules, instructed to use oral rinse, and received oral health education. Fixed orthodontic treatment with straight wire (AO self-ligating brackets, 0.022 x 0.028 inch slot, Empower® Philosophies, American Orthodontics, Sheboygan, USA) was used. The alignment and leveling procedures typically lasted three to four months. Subsequently, the orthodontic gap was closed by a 0.019 x 0.025 inch (0.48 mm x 0.64 mm) stainless steel square wire with a force gauge to control the sliding force value at approximately 150 g.

During orthodontic follow-up, the mobility of socket-shield, as well as clinical manifestations such as color, texture, and bleeding of gingiva, were evaluated to assess the clinical condition of the socket-shield.

2.3 Measurement methods In order to evaluate the clinical effects of SST and non-SST on alveolar bone width and height at the extraction site in the first premolar area, the left and right first premolars in same jaw were paired and randomly assigned to the test group (SST) or the control group (non-SST). The time points prior to tooth extraction, three months after tooth extraction, when the socket-shield extracted, and three months after socket-shield extraction were marked as T0, T1, T2, and T3 respectively. Cone beam computerized tomography (CBCT) scans (120 kVp and 18.66 mAs, voxel size 0.3, Alpha Plus RCT700-SC, RayScan, Hwaseong-si, Korea) were taken at each time point. T01 was defined as the interval from T0 to T1, T02 as T0 to T2, T12 as T1 to T2, T03 as T0 to T3, and T23 as T2 to T3.

Three-dimensional coordinate systems were established by CBCT data in Invivo Dental 5.0 software (Anatomage, Inc., Milan, Italy) to measure the alveolar bone height and width.

The most anterior-inferior point of the left mental foramen was defined as the origin, the line parallel to the line connecting the most anterior-inferior points of two mental foramina as the X-axis, and line parallel to the inferior border of the left mandible as the Y axes. Then, a three-dimensional coordinate system for the left mandible was established. A symmetric coordinate was established for the right mandible.

The most anterior point of the anterior nasal spine was set as the origin, the line parallel to the line connecting the lowest points of both maxillary sinus as the X-axis, and the line parallel to the palatal plane as Y-axis. Then, a three-dimensional coordinate system for the maxilla was established.

To ensure the consistency of the measurements at each time point, a cross-section parallel to the XZ plane through the lowest point of the alveolar crest was defined as the reference plane at T0. At T0, T1, T2, and T3, the Z value of the lowest point of the alveolar crest was recorded as alveolar bone height, and X value at 1 mm, 3 mm, and 5 mm from the reference plane was recorded as width, denoted as H0/W0(1,3,5), H1/W1(1,3,5), H2/W2(1,3,5), and H3/W3(1,3,5), respectively. The the changes of height and width can be calculated as follows: ΔH1=H1-H0/ΔW1=W1-W0 during T01, ΔH2=H2-H0/ΔW2=W2-W0 during T02, and ΔH3=H3-H0/ΔW3=W3-W0 during T03.

CBCT three-dimensional reconstruction graphics were used to measure the distance between the most convex points of the adjacent teeth in the mesial and distal distance of the orthodontic gap. Data at T1, T2, and T3 were recorded as D1, D2, and D3 respectively. Tooth movement rate can be calculated by dividing tooth movement distance (in mm) by the time taken for orthodontic gap closing (in months): (D1-D2)/(T2-T1) during T12 and (D2-D3)/(T3-T2) during T23.

All measurement were performed by two doctors who underwent standardized training. The data was subjected to a qualitative consistency test, the intraclass correlation coefficient (ICC). Only when ICC≥0.75, the average of the two measurements was used as the final result.

ELIGIBILITY:
Inclusion Criteria:

1. had an orthodontic treatment plan involving the extraction of symmetrical left and right first premolars;
2. had maxillary protrusion or bimaxillary protrusion with crowding within 4mm;
3. had permanent dentition;
4. had good oral hygiene and had no periodontitis;
5. agreed to the orthodontic extraction treatment plan and signed the treatment informed consent form and the experimental informed consent form.

Exclusion Criteria:

1. underlying diseases such as hypertension, heart disease, diabetes, osteoporosis, or hyperthyroidism;
2. infection in the extraction area;
3. dental root caries in the extraction area;
4. gingival recession on the buccal aspect of the extraction area;
5. refused to undergo SST treatments;
6. pregnancy or lactation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Vertical alveolar bone loss | 0 weeks, 3 months, 6 months and 9 months
  Cone beam computerized tomography were utilized to access the vertical resorption at 1mm, 3mm and 5mm from a reference plane of alveolar crest
Horizontal alveolar bone loss | 0 weeks, 3 months, 6 months and 9 months
  Cone beam computerized tomography were utilized to access the horizontal resorption at 1mm, 3mm and 5mm from a reference plane of alveolar crest

SECONDARY OUTCOMES:
Tooth movement rate | 3 months, 6 months and 9 months
  CBCT three-dimensional reconstruction graphics were used to measure the distance between the most convex points of the adjacent teeth in the mesial and distal distance of the orthodontic gap. Data at T1, T2, and T3 were recorded as D1, D2, and D3 respectively. Tooth movement rate can be calculated by dividing tooth movement distance (in mm) by the time taken for orthodontic gap closing (in months): (D1-D2)/(T2-T1) during T12 and (D2-D3)/(T3-T2) during T23.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxin Ji, DDS, Study Chair — The First Affiliated Hospital of Guangzhou Medical University; Yuhang Zhang, MS, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University; Zhe Ji, MS, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Ji Z, Lin L, Ye H, Ji J. The socket-shield technique in orthodontics: a method for alveolar ridge preservation. Oral Maxillofac Surg. 2026 Jan 10;30(1):16. doi: 10.1007/s10006-025-01501-9. PMID 41514150

DOCUMENTS (2):
  • Statistical Analysis Plan (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT06510621/SAP_000.pdf
  • Informed Consent Form (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT06510621/ICF_001.pdf